CLINICAL TRIAL: NCT01799590
Title: A Continuous Treatment Study of JNS019 (Topiramate) in Migraine Patients
Brief Title: Continuous Treatment Study of Topiramate in Migraine Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013684; JNS019-JPN-03
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Migraine
Keywords: Migraine; Topiramate
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate tablets will be administered orally in the dose range of 50 to100 milligram per day (mg/day). Dose will be increased or decreased as per Investigator's discretion. Maximum daily dose limit will be 200 mg.
  Other Names: JNS019

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of topiramate in participants with migraine (type of severe headache that occurs periodically and is often associated with nausea, vomiting and constipation or diarrhea) who completed the JNS019-JPN-02 study.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (conducted in more than one center), dose-titration (dose escalation/reduction) study of topiramate in participants with migraine. This study is a continuous study for the participants who were enrolled in the JNS019-JPN-02 study. Participants who completed the JNS019-JPN-02 study will receive treatment for 52 weeks starting at Visit 4 of the JNS019-JPN-02 study. The present study will consist of 3 weeks of Transfer period (during this period the dose titration will take place and along with dose titration the new treatment will be initiated at 25 milligram per day [25mg/day]), Continuous treatment period (32 weeks), Exit period (up to 3 weeks) and Follow-up period (4 weeks). Participants in the Continuous treatment period will receive topiramate tablets orally in the dose range of 50 mg/day to 100 mg/day. Dose can be increased or decreased as per Investigator's discretion. The maximum daily dose will be 200 mg/day. Efficacy will be primarily evaluated by change from Baseline in the number of monthly migraine attacks in Continuous treatment period. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- Participants who completed the JNS019-JPN-02 study or discontinued the study at Week 4 or after in fixed-dose period because of insufficient efficacy

Exclusion Criteria:

* Participants who discontinued the JNS019-JPN-02 study for an adverse event unrelated to the underlying disease
* Participants judged unfavorable to be transferred to this study because of the safety assessments in the JNS019-JPN-02 study
* Pregnant (carrying an unborn baby) female participants
* Other participants who were considered ineligible as per Investigator's discretion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (25):
- Japan (25):
  - Chitose
  - Hachiōji
  - Isehara
  - Kagoshima
  - Kamogawa
  - Kitakyushu
  - Kobe
  - Kumamoto
  - Kyoto
  - Minato
  - Morioka
  - Nagoya
  - Nishinomiya
  - Numakunai
  - Sagamihara
  - Sapporo
  - Shinjuku-Ku
  - Shizuoka
  - Suginami-Ku
  - Tokyo
  - Toyama
  - Toyonaka
  - Ube
  - Yokohama
  - Yonago

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Present study is continuation of previous study (JNS019-JPN-02, NCT01081795). The participants who completed the previous study or the cases where the administration of study drug was discontinued because of insufficient results were enrolled in this study.
Groups:
- Placebo/Topiramate (JNS019): Participants allocated to placebo group in the JNS019-JPN-02 trial were switched to active treatment in the current study JNS019-JPN-03. Participants received topiramate oral tablets twice daily in the dose range of 50 milligram (mg) to 100 mg. Dose was increased or decreased maximum up to 200 mg per day as per Investigators discretion. Total duration of treatment was 52 weeks.
- Topiramate (JNS019) 50 mg: Participants allocated to JNS019 50 mg group in JNS019-JPN-02 trial were switched to the dose range from 50 mg per day to 100 mg per day. Topiramate 25 mg oral tablets were administered twice daily. Dose was increased or decreased maximum up to 200 mg per day as per Investigators discretion. Total duration of treatment was 52 weeks.
- Topiramate (JNS019) 100 mg: Participants allocated to JNS019 100 mg group in JNS019-JPN-02 trial were switched to the dose range from 50 mg per day to 100 mg per day.Topiramate 50 mg oral tablets were administered twice daily. Dose was increased or decreased maximum up to 200 mg per day as per Investigators discretion. Total duration of treatment was 52 weeks.
Period: Overall Study
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Started | 111 | 94 | 91
Completed | 85 | 78 | 77
Not Completed | 26 | 16 | 14
Not completed — Adverse Event | 13 | 7 | 5
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 3
Not completed — Participants convenience | 4 | 4 | 2
Not completed — Aggravation of complications | 0 | 1 | 1
Not completed — Using drugs with restricted days of use | 0 | 3 | 2
Not completed — Use of prohibited concomitant drugs | 1 | 0 | 0
Not completed — Other | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg | Total
Number analyzed (Participants) | 111 | 94 | 91 | 296
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (8.83) | 40.7 (9.28) | 38.3 (9.12) | 40.3 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 74 | 66 | 232
  Male | 19 | 20 | 25 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Baseline up to 28 days after last dose of study drug
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Participants | 110 | 85 | 79

2. Secondary Outcome: Change From Baseline in the Number of Monthly Migraine Attacks as Per 24-hour Rule in the Continuous Treatment Period
Description: As per 24-hour rule, if symptom of pain because of migraine continues for more than 24 hours, it should be considered as 2 or more migraine attacks considering the maximum duration up to 24 hours. If interval between the latest migraine attack (ending time) and previous migraine attack (onset time) was less than 24 hours, 2 migraine attacks were considered as 1 migraine attack. If the onset of the migraine was prevented by a rescue drug it was considered as 1 migraine attack even if the aura had started.
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: Full analysis set (FAS) included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization.
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Migraine attacks
  Baseline (28 days before randomization) | 6.5 (2.27) | 5.9 (1.76) | 6.0 (1.91)
  Change during Continuous treatment period | -2.1 (2.47) | -1.0 (3.21) | -1.6 (2.11)

3. Secondary Outcome: Change From Baseline in the Average Number of Monthly Migraine Attack Days in Continuous Treatment Period
Description: Migraine:disabling headache disorder;2 major subtypes:migraine without aura(at least 5 attacks for 4-72 hours with at least 2 characteristics: unilateral location,pulsating quality,moderate/severe pain intensity or aggravation by/causing avoidance of routine physical activity and either nausea/vomiting or photophobia,phonophobia);migraine with aura(attack with reversible focal neurological symptoms that develop over 5-20 minutes, last for less than 60 minutes);average=total number of migraine attack days divided by total number of days of assessment and multiplied by 28,where a month=28 days.
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: The FAS included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Days
  Baseline (28 days before randomization) | 7.3 (2.56) | 6.5 (2.09) | 6.7 (2.16)
  Change during Continuous treatment period | -2.4 (2.78) | -1.1 (3.24) | -1.9 (2.44)

4. Secondary Outcome: Change From Baseline in the Average Number of Monthly Headache Days in Continuous Treatment Period
Description: Migraine headache day was defined as a calendar day with any occurrence of migraine headache pain of at least 30 minutes in duration. Average was calculated as total number of monthly headache days divided by total number of days of assessment and multiplied by 28, where a month was considered to last 28 days.
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Days
  Baseline (28 days before randomization) | 7.5 (2.73) | 6.8 (2.07) | 7.2 (2.36)
  Change during Continuous treatment period | -2.6 (2.75) | -1.2 (3.28) | -2.1 (2.52)

5. Secondary Outcome: Change From Baseline in the Average Number of Migraine Attacks According to the Diagnostic Criteria of the International Headache Society Per Month in Continuous Treatment Period
Description: Migraine has 2 major subtypes: migraine without aura (minimum 5 attacks of headache lasting for 4-72 hours, has 2 of these characteristics [unilateral location, pulsating quality, moderate or severe pain intensity, aggravation by or causing avoidance of routine physical activity] and either nausea/vomiting or photophobia and phonophobia) and migraine with aura (2 attacks of headache with typical aura with migraine headache or typical aura with non-migraine headache or typical aura without headache or familial hemiplegic migraine or sporadic hemiplegic migraine or basilar-type migraine).
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Migraine attacks
  Baseline (28 days before randomization) | 4.7 (2.94) | 4.6 (2.33) | 4.6 (2.89)
  Change during Continuous treatment period | -1.9 (2.39) | -1.6 (2.40) | -1.6 (2.25)

6. Secondary Outcome: Change From Baseline in the Number of Monthly Migraine Attacks as Per 48-hour Rule in Continuous Treatment Period
Description: As per 48-hour rule, if the symptom of pain because of migraine continues for more than 48 hours, it should be considered as 2 or more migraine attacks considering the maximum duration up to 48 hours. If the interval between the latest migraine attack (ending time) and the previous migraine attack (onset time) is less than 48 hours, 2 migraine attacks were considered as 1 migraine attack. If the onset of the migraine was prevented by a rescue drug it was considered as 1 migraine attack even if the aura had started.
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Migraine attacks
  Baseline (28 days before randomization) | 5.0 (1.58) | 4.6 (1.23) | 4.8 (1.41)
  Change during Continuous treatment period | -1.6 (1.76) | -0.9 (1.91) | -1.3 (1.60)

7. Secondary Outcome: Change From Baseline in the Number of Migraine Attacks as Per 24-hour Rule Over Day 197 to Day 225 in Continuous Treatment Period
Description: As per 24-hour rule, if symptom of pain because of migraine continues for more than 24 hours, it should be considered as 2 or more migraine attacks considering the maximum duration up to 24 hours. If interval between the latest migraine attack (ending time) and previous migraine attack (onset time) is less than 24 hours, 2 migraine attacks were considered as 1 migraine attack. If the onset of the migraine was prevented by a rescue drug it was considered as 1 migraine attack even if the aura had started.
Time Frame: Baseline (28 days before randomization) and Day 197 to Day 225
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Migraine attacks
  Baseline (28 days before randomization) | 6.5 (2.27) | 5.9 (1.76) | 6.0 (1.91)
  Change during Day 197 to 225 | -1.9 (2.87) | -1.1 (3.33) | -1.4 (2.68)

8. Secondary Outcome: Change From Baseline in the Average Number of Monthly Rescue-Drug Treatment Days in Continuous Treatment Period
Description: If aura of migraine, migraine attack or non-migraine headache attack occurred in study, these rescue drugs were permitted:analgesics, non-steroidal anti-inflammatory drugs (NSAIDs),ergotamines,triptans,antiemetics. Drugs with restricted treatment days of less than (<) 15 days per month (28 days):analgesics, NSAIDs,combination of rescue drugs and those with <10 days per month:triptans,ergotamines, opioids,combination analgesics. Average calculated as total number of monthly rescue-drug treatment days divided by the total number of days of assessment and multiplied by 28, where a month = 28 days.
Time Frame: Baseline (28 days before randomization) and Continuous treatment period (Day 1 up to Day 225)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Days
  Baseline (28 days before randomization) | 5.9 (2.35) | 5.5 (2.21) | 5.2 (2.26)
  Change during Continuous treatment period | -1.6 (2.43) | -0.7 (3.08) | -1.0 (2.16)

9. Secondary Outcome: Percentage of Participants With Response to Treatment
Description: Responders were defined as participants who had a 50 percent or more reduction in frequency of migraine attacks. Migraine is common disabling headache disorder with 2 subtypes: migraine without aura (at least 5 attacks lasting 4-72 hours with at least 2 characteristics: unilateral location, pulsating quality, moderate/severe pain or aggravation by/causing avoidance of routine physical activity and either nausea/vomiting or photophobia and phonophobia) and migraine with aura (attack with reversible focal neurological symptoms that develop over 5-20 minutes and last for less than 60 minutes).
Time Frame: Baseline (28 days before randomization) up to Day 225
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Percentage of participants | 36.0 | 18.1 | 22.0

10. Secondary Outcome: Quality of Life (QOL) Questionnaire (Short Form-36 [SF-36]) Score
Description: The SF-36 is a standardized survey evaluating 8 domains (consisting of 2 components; physical and mental) of functional health and well being: physical and social functioning, physical and emotional role (role-physical, role-emotional) limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Final evaluation (FE) was done at Day 225 or at discontinuation.
Time Frame: Baseline (28 days before randomization) and FE (Day 225/early discontinuation)
Population: The FAS included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization. Here 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Number analyzed (Participants) | 111 | 94 | 91
Units on a scale
  Body function: Baseline (n=111,94,91) | 54.06 (5.957) | 53.52 (5.033) | 54.10 (8.374)
  Body function: FE (n=109,89,91) | 53.14 (8.269) | 54.35 (5.648) | 54.79 (6.184)
  Daily activity (physical): Baseline (n=111,94,91) | 45.81 (9.556) | 45.45 (9.909) | 46.15 (10.916)
  Daily activity (physical): FE (n=109,89,91) | 45.50 (11.220) | 45.96 (9.789) | 47.34 (9.804)
  Body pain: Baseline (n=111,94,91) | 39.90 (9.496) | 41.06 (8.274) | 42.77 (10.549)
  Body pain: FE (n=109,89,91) | 43.07 (9.744) | 43.95 (10.725) | 43.87 (9.861)
  Overall health: Baseline (n=111,94,91) | 48.01 (7.526) | 47.65 (8.895) | 49.39 (8.413)
  Overall health: FE (n=109,89,91) | 49.75 (9.373) | 47.07 (9.564) | 50.72 (9.622)
  Energy: Baseline (n=111,94,91) | 49.43 (8.392) | 48.73 (7.849) | 49.84 (7.269)
  Energy: FE (n=109,89,91) | 48.85 (9.468) | 48.10 (9.796) | 48.18 (9.644)
  Social activities: Baseline (n=111,94,91) | 47.49 (10.373) | 47.71 (9.959) | 49.07 (9.891)
  Social activities: FE (n=109,89,91) | 46.23 (11.405) | 46.74 (10.349) | 50.22 (8.318)
  Daily activity (mental): Baseline (n=111,94,91) | 51.23 (8.862) | 51.34 (7.879) | 51.36 (8.990)
  Daily activity (mental): FE (n=109,89,91) | 48.59 (10.273) | 48.51 (9.271) | 49.53 (9.173)
  Mental health: Baseline (n=111,94,91) | 50.95 (8.728) | 50.55 (8.017) | 50.80 (7.958)
  Mental health: FE (n=109,89,91) | 48.16 (9.836) | 47.86 (9.514) | 49.64 (9.801)
  Physical component summary: Baseline (n=111,94,91) | 48.37 (7.425) | 48.42 (7.497) | 49.05 (9.455)
  Physical component summary: FE (n=109,89,91) | 48.10 (9.989) | 49.22 (8.982) | 50.17 (7.718)
  Mental component summary: Baseline (n=111,94,91) | 48.3 (7.923) | 48.06 (7.682) | 49.23 (7.383)
  Mental component summary : FE (n=109,89,91) | 47.73 (9.471) | 46.49 (46.49) | 48.36 (9.087)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug
Arm/Group | Placebo/Topiramate (JNS019) | Topiramate (JNS019) 50 mg | Topiramate (JNS019) 100 mg
Serious Adverse Events (participants affected / at risk) | 3/111 | 0/94 | 2/91
Other Adverse Events (participants affected / at risk) | 110/111 | 85/94 | 79/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Topiramate (JNS019) (N=111) | Topiramate (JNS019) 50 mg (N=94) | Topiramate (JNS019) 100 mg (N=91)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Topiramate (JNS019) (N=111) | Topiramate (JNS019) 50 mg (N=94) | Topiramate (JNS019) 100 mg (N=91)
Nasopharyngitis (Infections and infestations) | 39 | 36 | 36
Gastroenteritis (Infections and infestations) | 8 | 5 | 4
Cystitis (Infections and infestations) | 6 | 3 | 3
Influenza (Infections and infestations) | 2 | 1 | 6
Seasonal allergy (Immune system disorders) | 7 | 5 | 3
Loss of appetite (Metabolism and nutrition disorders) | 12 | 4 | 5
Dysesthesia (Nervous system disorders) | 42 | 15 | 11
Paraesthesia (Nervous system disorders) | 32 | 12 | 8
Drowsiness (Nervous system disorders) | 11 | 6 | 7
Dizziness (Nervous system disorders) | 4 | 1 | 8
Neuralgia (Nervous system disorders) | 8 | 1 | 0
Inflammation of upper respiratory tract (Respiratory, thoracic and mediastinal disorders) | 14 | 12 | 14
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 1
Diarrhea (Gastrointestinal disorders) | 15 | 3 | 4
Gastritis (Gastrointestinal disorders) | 8 | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 6 | 5 | 5
Nausea (Gastrointestinal disorders) | 6 | 5 | 1
Constipation (Gastrointestinal disorders) | 6 | 2 | 1
Decayed tooth (Gastrointestinal disorders) | 1 | 5 | 2
Backache (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 | 2 | 1
Fatigue (General disorders) | 13 | 3 | 3
Laboratory tests (General disorders) | 73 | 48 | 42
Weight reduction (General disorders) | 57 | 36 | 29
Decrease blood bicarbonate (General disorders) | 20 | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the Sponsor requires.